CLINICAL TRIAL: NCT03759860
Title: A Prospective, Single-Center, Randomized, Double Blind, Double Arm, Comparative Clinical Trial to Compare the Safety and Preliminary Efficacy Between Ranibizumab Monotherapy and Ranibizumab Combined With R:GEN (Selective Retina Therapy) in Clinically Significant Diabetic Macular Edema (a Pilot Study)
Brief Title: Laser (Selective Retina Therapy) and Drug Combined Intervention in Clinically Significant Diabetic Macular Edema
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CynosureLutronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSDME_P01
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab; Combined Modality Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant must be masked from the information on the treatment group assignment.
  The BCVA and image (OCT, Color Fundus Photography (CFP), Fundus Autofluorescence (FAF), Fluorescence Angiography (FAG)) investigator of the institution must be blinded on the participants' treatment group assignment to eliminate bias in evaluation.
  Based on the images (OCT, CFP, FAF) and quantified measurement results (BCVA, OCT), the blinded principal investigator (independent evaluator) evaluates efficacy and adverse events and determines whether ranibizumab should be administered again.
  An investigator not blinded performs SRT and ranibizumab administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Selective Retina Therapy and ranibizumab combination therapy (Experimental): Perform R:GEN laser (SRT) on the 6,000 microns diameter region including macular edema, while excluding the 500 microns diameter region from the fovea, with the appropriate treatment energy determined.
  Ranibizumab (Lucentis®; Novartis AG, Basel, Switzerland) injection into the vitreous cavity at 3.5-4.0 mm posterior to the corneal limbus, towards the center of the eye, avoiding horizontal meridians. Then, 0.05 mL of the injection solution is slowly injected.
  In study group and the control group, ranibizumab is administered 5 times in total from the baseline to month 4.
  Interventions: Combination Product: R:GEN laser treatment (Selective Retina Therapy) and Lucentis (ranibizumab) combination therapy
- Sham Selective Retina Therapy and ranibizumab monotherapy (Sham Comparator): For the participants assigned to the control group, sham procedures are performed in Sham Mode. All procedures except for the absence of laser light emission at the laser irradiation stage are the same with the study group.
  Sham SRT is performed three times in total, one time for each visit for month 1, 3, and 5. At the time of month 1 and 3, Sham SRT should be performed before administration of ranibizumab.
  Interventions: Combination Product: R:GEN laser treatment (Selective Retina Therapy) and Lucentis (ranibizumab) combination therapy

INTERVENTIONS:
Combination Product: R:GEN laser treatment (Selective Retina Therapy) and Lucentis (ranibizumab) combination therapy — Lucentis (ranibizumab) injection into the vitreous cavity after R:GEN laser treatment (Selective Retina Therapy)

SUMMARY:
The objective of this clinical trial is to compare and evaluate the safety and efficacy of Ranibizumab (Lucentis®; Novartis AG, Basel, Switzerland) monotherapy and Ranibizumab combined with R:GEN (Selective Retina Therapy) in patients with clinically significant diabetic macular edema.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized, double blind, double arm, comparative clinical trial to compare the safety and efficacy between ranibizumab monotherapy and ranibizumab combined with Selective Retina Therapy (SRT) in clinically significant diabetic macular edema (a pilot study).

Screening visit should be conducted within 30 days before the baseline visit. After assigning a screening number (SN) to the participants who voluntarily agreed in writing to participate in the clinical trial, conduct a screening test to determine whether the subject meet the inclusion/ exclusion criteria.

Proceed with the clinical trial with the appropriate subjects determined based on the inclusion/exclusion criteria. Random allocation numbers (AN) are assigned.

Participants are randomly assigned to study group or control group. Combination therapy of SRT and ranibizumab is performed in the study group and sham SRT and ranibizumab monotherapy is performed in the control group. (Sham) SRT and ranibizumab (re-performance) is performed by the institution's investigator other than the independent evaluator.

In the study group and control group, after the completion of 5 ranibizumab injections during the loading period, if the independent evaluator judges the following criteria apply based on Best Corrected Visual Acuity (BCVA) and Optical Coherence Tomography (OCT) findings at each visit from the 5th month, ranibizumab is re-administered by an investigator other than the independent evaluator, within 14 days of the visit or on the day of visit; If the independent evaluator judges that CMT on the OCT is equal to or greater than the baseline; or if the independent evaluator judges that BCVA is equal to or worse than the baseline.

The study group and the control group visit the hospital at the time of (Sham) SRT and ranibizumab performance from the baseline until 5 months and make a visit every month from 6 months to 12 months.

From 13 months ± 14 days after the baseline, the schedule of visits can be determined at intervals of 1 month ± 14 days to 3 months ± 14 days at the discretion of the investigator other than the independent evaluator. However, at the time of 24 months, both the study group and the control group should visit the hospital for efficacy and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults older than 19 years of age
2. Patients with Type-I or Type-II diabetes
3. Patients diagnosed with Clinically Significant Diabetic macular edema (CSME) based on the criteria of Early Treatment Diabetic Retinopathy Study (ETDRS).

   * If thickened retina is within or lies on the circle with a radius of 500µm from the center of the fovea, or
   * If the hard exudate is within or lies on the circle with a radius of 500 ㎛ and if the retina adjacent to it is thickened, or
   * If there is a thickened retina larger than 1 disc area and if a part of it is over the circle with a radius of 1 disc diameter from the center of the macula.
4. Central Macular Thickness (CMT) of study eye is more than 300㎛ on OCT
5. Patients with BCVA of the study eye between 20/320 and 20/25.
6. Patients who have agreed to participate in this study and signed the consent form, and patients whose legally acceptable representative signed the consent form

Exclusion Criteria:

1. Patients with Ischemic DME that showed rupture in the Foveal Avascular Zone due to the obstruction of more than 30% of the capillary vessels in the central circle, as observed using fluorescein angiography
2. Patients with a history of focal steroid treatment in the study eye within 4 months
3. Patients with a history of anti-VEGF agent injection in the study eye within 3 months
4. Patients with rubeosis iridis, vitreous hemorrhage or tractional retinal detachment in the study eye
5. Patients with uncontrolled glaucoma in the study eye
6. Patients with active inflammation or infection in the study eye (in or around the eye)
7. Patients with disorders in the study eye that may confuse interpretation of the clinical trial results, cause severe visual loss, and require medical or surgical intervention during the study, based on the investigator's judgment (media opacity such as corneal opacity, cataract, and vitreous opacity, vitreous macular traction, uveitis, macular atrophy, macular degeneration, choroidal neovascularization, retinal vascular occlusion)
8. Persons with a history of treatment with anti-VEGF drugs within the past 6 months, or if they anticipate future use (e.g.: sorafenib (Nexavar®), sunitinib (Sutent®), bevacizumab (Avastin®))
9. Persons with confirmed allergy to fluorescein, indocyanine green or iodine
10. Patients with a clinically significant disorder such as uncontrolled renal failure that would make it difficult for them to participate in this study, based on the investigator's judgment
11. Pregnant or lactating woman
12. Patient not using contraception or with a possibility of pregnancy during the clinical trial period
13. Other persons deemed to be difficult to participate in this study, based on the investigator's judgment
14. Persons participating in a study other than observational or non-interventional study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) change in the study group | 12 months
  Compare BCVA change evaluated between the group where Ranibizumab was combined with R:GEN (Selective Retina Therapy) and the group where Ranibizumab monotherapy was applied

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) change in the study group | 12, 24 months
  Compare BCVA change evaluated between the group where Ranibizumab was combined with R:GEN (Selective Retina Therapy) and the group where Ranibizumab monotherapy was applied
Central Macular Thickness (CMT) change in the study group | 12, 24 months
  Compare CMT change evaluated between the group where Ranibizumab was combined with R:GEN (SRT) and the group where Ranibizumab monotherapy was applied.
Maximum Macular Thickness (MMT) change in the study group | 12, 24 months
  Compare MMT change evaluated between the group where Ranibizumab was combined with R:GEN (SRT) and the group where Ranibizumab monotherapy was applied.
Rate and number of Ranibizumab re-performance in the study group | 24 months
  Compare the rate of participants who received Ranibizumab re-performance and the number of Ranibizumab re-performance between the group where Ranibizumab was combined with R:GEN (SRT) and the group where Ranibizumab monotherapy was applied.
Adverse Event analysis | 24 months
  Evaluate safety by comparing the rate of participants who experienced Adverse Event.

CONTACTS AND LOCATIONS:
Overall Officials: Hakyung Kim, Professor, Principal Investigator — Hallym University Kangnam Sacred Heart Hospital
Locations (1):
- Hallym University Kangnam Sacred Heart Hospital, Seoul, South Korea